CLINICAL TRIAL: NCT03606629
Title: Solaris Endoprosthesis Performance in Treatment of Patients With Peripheral Occlusive Arterial Disease in the Iliac Territory - Post-Marketing Solaris I Study.
Brief Title: SOLARIS Endoprosthesis in Iliac Occlusive Disease
Acronym: SOLARIS I
Status: Completed | Type: Observational
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: SC-SO-001
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoprosthesis implantation: Device implantation
  Interventions: Device: Endoprosthesis implantation

INTERVENTIONS:
Device: Endoprosthesis implantation — Endoprosthesis implantation by Percutaneous Angioplasty

SUMMARY:
Fifty patients will be treated with Solaris Endoprosthesis and followed up to 2 years with Walking Impairment Questionnaire and Doppler Ultrasound evaluation in 30 days, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford Class 2 to 5;
* Tasc II Class A, B, C or D;
* Unilateral or bilateral lesion, de novo or restenotic but not in-stent;
* Target lesion of 3 to 10 cm length;
* ≥ 50% stenosis or common iliac or external iliac artery;
* Reference vessel diameter ≥ 5 and ≤ 9 mm;
* Deep femoral artery patent and at least one infrapopliteal artery patent;
* Informed Consent provided.

Exclusion Criteria:

* Thrombocytopenia induced by heparina or tPA intravenous, clopidogrel, ticlopidine or aspirin sensitivity;
* Target lesion near to aneurysm, highly calcified or excessively tortuous;
* Previous stent on target vessel;
* Presence of other lesions that need treatment within 30 days;
* Rutherford Class 6;
* Acute thrombotic occlusion;
* History on amputation on the target limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with POAD presenting limitant intermitent claudication after 6 months of clinical treatment and patients with rest ischemia, Rutherford class 2 to 5.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Events | 1 day
  MAE is defined as death related to study device/ procedure, Myocardial Infarction, Target Vessel Revascularization or member amputation
Target Lesion Patency | 6 months
  Stenosis < 50% and systolic velocity up to 2.5 cm2/s and no TLR

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Furuya, MD, Principal Investigator — Santa Casa de Misericórdia de Santo Amaro
Locations (1):
- Hospital de Clínicas de Passo Fundo, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No